CLINICAL TRIAL: NCT05174429
Title: Risk-Targeted Behavioral Activation for the Management of Work-Disability Associated With Co-Morbid Pain and Depression: A Feasibility Study
Brief Title: The Management of Work-Disability Associated With Co-Morbid Pain and Depression: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: l'Institut de recherche Robert-Sauvé en santé et en sécurité du travail (IRSST) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0024
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Risk-Targeted Behavioral Activation (Experimental): The treatment program consisted of a 10-week standardized behavioral activation intervention supplemented by techniques to target two psychosocial risk-factors for delayed recovery, namely, catastrophic thinking and perceptions of injustice.
  Interventions: Behavioral: Risk-Targeted Behavioral Activation

INTERVENTIONS:
Behavioral: Risk-Targeted Behavioral Activation — The behavioral activation component of the treatment program focused on goal setting, structuring and scheduling activities, increasing success and achievement experiences, and problem-solving. In order to maximize the impact of behavioral activation on disability reduction, goal setting and scheduling of activities focused primarily on resumption of discontinued activities as opposed to focusing on the scheduling of pleasant activities. One objective of goal setting and activity scheduling was to reduce the discrepancy between the client's pre-injury activity repertoire and the client's current activity repertoire.
  Behavioral activation was supplemented by a collection of techniques designed to reduce catastrophic thinking and perceptions of injustice, two psychosocial risk factors that have been shown to contribute to prolonged work-absence.

SUMMARY:
The purpose of the present study was to conduct a preliminary evaluation the feasibility and impact of a risk-targeted behavioral activation intervention for work-disabled individuals with co-morbid pain and depression.

DETAILED DESCRIPTION:
The design of the study was a single arm non-randomized trial. The sample consisted of 66 work-disabled individuals with co-morbid pain and depression. The treatment program consisted of a 10-week standardized behavioral activation intervention supplemented by techniques to target two psychosocial risk-factors for delayed recovery, namely, catastrophic thinking and perceptions of injustice.

ELIGIBILITY:
Inclusion Criteria:

* 1) work-disability greater than 4 weeks associated with a musculoskeletal injury to the back or neck, 2) a score above clinical threshold on a self-report measure of depression, and 3) between 25 and 55 years of age.

Exclusion Criteria:

* 1) Clinical evidence of vertebral fracture, disk herniation, infectious disease, or rheumatoid arthritis: 2) Evidence of chronic pain pre-dating the current injury: 3) Evidence of loss of consciousness at the time of injury: 4) Previous musculoskeletal injury sustained within the past 12 months: 5) Evidence of any medical condition that might contraindicate participation in physical activity: 6) Illiteracy or severe cognitive impairment.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Return to work | Assessed 6 months following termination of treatment.
  Percentage of participants who resumed employment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sullivan, PhD, Principal Investigator — McGill University

IPD SHARING:
Plan to Share IPD: No